CLINICAL TRIAL: NCT00001993
Title: Initial Phase II Efficacy and Safety Study of SC-48334 Administered in Combination With Low-Dose Zidovudine (AZT) to Symptomatic HIV-1 Infected Patients With = or > 200 to = or < 500 CD4+ Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G D Searle (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 057A; NS8-90-02-004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — miglustat; Zidovudine

INTERVENTIONS:
Drug: Butyldeoxynojirimycin
Drug: Zidovudine

SUMMARY:
The primary objective of this study is to determine the preliminary efficacy and tolerability of combining a selected dose of SC-48334 with low-dose AZT in the treatment of symptomatic HIV+ patients with 200 to 500 CD4+ cells/mm3.

The secondary objective is to determine the pharmacokinetics and bioavailability of both SC-48334 and AZT, when administered together, in symptomatic HIV+ patients with 200 - 500 CD4+ cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Medications for the prophylaxis of opportunistic infections, such as:
* Aerosolized pentamidine.
* Trimethoprim/sulfamethoxazole.
* Nystatin.
* Clotrimazole.
* Anti-mycobacterial agents.
* Ganciclovir.
* Topical acyclovir.

Patients must have the following:

* CD4+ cells counts = or > 200 < 500 /cell mm3.
* For purposes of inclusion the absolute CD4+ cell count must be = or > 200 < 500 cells/mm3 on the first sample and = or > 190 < 510 cells/mm3 on the second sample.
* Have at least one of the following:
* Oral candidiasis.
* Herpes zoster during the last 3 years.
* Oral hairy leukoplakia during the past three years.
* Chronic ( > 30 day period), recurrent seborrheic dermatitis, or topical, pruritic folliculitis (itchy bumps).
* Unintentional weight loss in excess of 10 pounds or 10 percent of usual body weight.
* Chronic fatigue present for the past 6 months, which has interfered with normal activity at least 1 to 2 times per week.
* HIV antibody positive as determined by federally licensed Enzyme-linked Immunosorbent Assay (ELISA).
* Documented, written informed consent must be obtained prior to admission to the study.

Prior Medication:

Allowed for no more than 12 weeks prior to study entry:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malignancies, with the exception of basal cell carcinoma.
* Significant organ dysfunction.

Concurrent Medication:

Excluded:

* All anti-retroviral drugs with the exception of Zidovudine. Cancer chemotherapeutic agents.
* Anti-metabolites and alkylating agents.
* All investigational non-FDA approved drugs.

Patients with the following are excluded:

* Clinically significant diarrhea (> 3 liquid stools per day for > 7 days) without definable cause, within 6 months prior to enrollment).
* Diarrhea, as above, with known, non-HIV related cause occurring within one month prior to enrollment.
* Meets CDC criteria for AIDS classification.
* Chronic fever (> 38.5 C persisting for more than 14 consecutive days, or for more than 15 days in any 30-day interval prior to study entry).
* Malignancies, with the exception of basal cell carcinoma.
* Significant organ dysfunction.
* Known hypersensitivity to SC-48334 or related compounds.
* History of lactose intolerance.

Prior Medication:

Excluded within 30 days of study entry:

* Any investigational medication.
* Treatment with a drug (other than Zidovudine) with anti-HIV activity.
* Excluded for > 12 weeks prior to study entry:
* Zidovudine (AZT).
* Excluded within 90 days of study entry:
* Ribavirin.
* Excluded within 6 months of study entry:
* Cancer chemotherapy.
* Excluded:
* Treatment with SC-48334.

Prior Treatment:

Excluded within 30 days of study entry:

* Electron beam radiation.
* Excluded within 6 months prior to study entry:
* Required HIV-related blood transfusions.
* Whole body radiation.

Current use of illicit substances; or current abuse of alcohol, the use of which would limit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Univ of Miami School of Medicine, Miami, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Fischl MA, Resnick L, Coombs R, Kremer AB, Pottage JC Jr, Fass RJ, Fife KH, Powderly WG, Collier AC, Aspinall RL, et al. The safety and efficacy of combination N-butyl-deoxynojirimycin (SC-48334) and zidovudine in patients with HIV-1 infection and 200-500 CD4 cells/mm3. J Acquir Immune Defic Syndr (1988). 1994 Feb;7(2):139-47. PMID 7905523